CLINICAL TRIAL: NCT03891953
Title: A Phase I/Ib, Open-label, Multi-center, Study of DKY709 as a Single Agent and in Combination With PDR001 in Patients With Advanced Solid Tumors
Brief Title: Study of Safety and Efficacy of DKY709 Alone or in Combination With PDR001 in Patients With Advanced Solid Tumors.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDKY709A12101C; 2018-002580-26 (EudraCT Number)
Record Dates: First submitted 2019-03-26; First posted 2019-03-27 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Melanoma; Nasopharyngeal Carcinoma; Microsatellite Stable Colorectal Cancer; Triple Negative Breast Cancer
Keywords: Non-small Cell Lung Cancer; Melanoma; Nasopharyngeal Carcinoma; Microsatellite Stable Colorectal Cancer; Triple Negative Breast Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Nasopharyngeal Carcinoma; Triple Negative Breast Neoplasms | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DKY709 (Experimental): DKY709 monotherapy
  Interventions: Drug: DKY709
- DKY709 + PDR001 (Experimental): Combination therapy with DKY709 and PDR001
  Interventions: Drug: DKY709; Drug: PDR001

INTERVENTIONS:
Drug: DKY709 — Novel immunomodulatory agent
Drug: PDR001 — PDR001 is a high-affinity, ligand-blocking, humanized IgG4 monoclonal antibody directed against PD-1 that blocks the binding of PD-L1 and PD-L2
  Other Names: Spartalizumab
  Arms: DKY709 + PDR001

SUMMARY:
This is a phase I/Ib, open label study. The escalation portion will characterize the safety and tolerability of DKY709 and DKY709 in combination with PDR001 in subjects with NSCLC or melanoma who have received prior anti-PD-1/PD-L1 therapy, or subjects with NPC. After the determination of the MTD/RD for a particular treatment arm, dose expansion will further assess safety, tolerability, PK/PD, and anti-tumor activity of each regimen at the MTD/RD.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study.
2. Patients must be ≥18 years of age at the time of informed consent form (ICF) signature.
3. Patients with advanced/metastatic cancer who have progressed despite having received standard therapy in the metastatic setting or are intolerant to standard therapy, and for whom no effective standard therapy is available
4. In expansion: patient with measurable disease as determined by RECIST version 1.1,
5. Dose escalation, patients must fit into one of the following groups:

   * NSCLC, previously treated with an anti-PD-1/PD-L1 therapy
   * Cutaneous Melanoma, previously treated with an anti-PD-1/PD-L1 therapy
   * NPC

   Dose expansion part, patients must fit into one of the following groups:
   * NSCLC with historic documentation of PD-L1 ≥ 1%. Patients must have progressive disease after having experienced at least 4 months of investigator-assessed disease stability or response on prior anti-PD-L1-containing therapy
   * Cutaneous Melanoma, previously treated with anit-PD-1/PD-L1 therapy. Patients should have documented progression following anti-PD-1/PD-L1 therapy.
   * NPC, naive to anti-PD-1/PD-L1 therapy
   * mssCRC, naive to anti-PD-1/PD-L1 therapy
   * TNBC, naive to anti-PD-1/PD-L1 therapy
6. ECOG Performance Status ≤ 1
7. Patients must have a site of disease amenable to core needle biopsy, and be a candidate for tumor biopsy according to the treating institution's guidelines. Patients must be willing to undergo a new tumor biopsy at baseline, and during therapy on the study. Exceptions may be considered after documented discussion with Novartis.

Exclusion Criteria:

1. Presence of symptomatic central nervous system (CNS) metastases, or CNS metastases that require local CNS-directed therapy (such as radiotherapy or surgery), or increasing doses of corticosteroids within 2 weeks prior to study entry. Patients with treated brain metastases should be neurologically stable for at least 4 weeks prior to study entry and off steroids for at least 2 weeks before administration of any study treatment.
2. History of severe hypersensitivity reactions to any ingredient of study drug(s) or other mAbs and/or their excipients.
3. Patient with out of range laboratory values defined as:

   * Creatinine clearance (calculated using Cockcroft-Gault formula, or measured) < 40 mL/min
   * Total bilirubin > 1.5 x ULN, except for patients with Gilbert's syndrome who are excluded if total bilirubin > 3.0 x ULN or direct bilirubin > 1.5 x ULN
   * Alanine aminotransferase (ALT) > 3 x ULN, except for patients that have tumor involvement of the liver, who are excluded if ALT > 5 x ULN
   * Aspartate aminotransferase (AST) > 3 x ULN, except for patients that have tumor involvement of the liver, who are excluded if AST > 5 x ULN
   * Absolute neutrophil count (ANC) < 1.0 x 109/L
   * Platelet count < 75 x 109/L (growth factor or transfusion support may not be used to meet entry criterion)
   * Hemoglobin (Hgb) < 8 g/dL (growth factor or transfusion support may not be used to meet entry criterion)
   * Magnesium, calcium or phosphate abnormality CTCAE > grade 1
   * Potassium abnormality CTCAE ≥ grade 1; supplementation to meet eligibility criteria is acceptable
4. Clinically significant cardiac disease or impaired cardiac function, including any of the following:

   * Clinically significant and/or uncontrolled heart disease such as congestive heart failure requiring treatment (NYHA grade ≥ 2), uncontrolled hypertension or clinically significant arrhythmia
   * On screening: QTcF > 450 msec (male), or > 460 msec (female)
   * QTc not assessable
   * Congenital long QT syndrome
   * History of familial long QT syndrome or known family history of as Torsades de Pointes
   * Acute myocardial infarction or unstable angina pectoris < 3 months prior to study entry

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Safety of DKY709 single agent treatment or DKY709 in combination with PDR001. | 24 months
  Incidence and severity of AEs and SAEs
incidence of Dose Limiting Toxicities (DLTs) | 1 Month
  The incidence of DLTs during the first cycle of treatment with single agent DKY709 or the combination of DKY709 with PDR001.
Tolerability of DKY709 single agent treatment or DKY709 in combination with PDR001. | 24 months
  Incidence and severity of AEs and SAEs

SECONDARY OUTCOMES:
AUC of DKY709 and PDR001 | 24 months
  AUC
Cmax of DKY709 and PDR001 | 24 months
  Cmax
Tmax of DKY709 and PDR001 | 24 months
  Tmax
Half-life of DKY709 and PDR001 | 24 months
  Half-life
Progression Free Survival (PFS) | 24 months
  Determine PFS in each part of the study
Best Overall Response (BOR) | 24 months
  Determine BOR in each part of the study
Duration of Response (DOR) | 24 months
  Determine DOR in each part of the study
Time to Progression (TTP) | 24 months
  Determine TTP in each part of the study

CONTACTS AND LOCATIONS:
Locations (9):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Germany (2):
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Essen
- Novartis Investigative Site, Hong Kong, Hong Kong
- Novartis Investigative Site, Chuo Ku, Tokyo, Japan
- Novartis Investigative Site, Barcelona, Spain
- Novartis Investigative Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No